CLINICAL TRIAL: NCT03488862
Title: Pilot Evaluation of a Microfluidic Assay to Detect Minimal Residual Disease and Predict Relapse in Acute Myeloid Leukemia (AML) Patients in Remission Following Allogeneic Stem Cell Transplant or Induction and Consolidation Chemotherapy
Brief Title: Pilot Evaluation of a Microfluidic Assay to Detect Minimal Residual Disease and Predict Relapse in AML Patients
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC 1702
Record Dates: First submitted 2018-03-28; First posted 2018-04-05 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Residual blood samples may be stored by the sponsor as backup to be used to confirm downstream assays using staining, fluorescence-activated cell sorting (FACS).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Purpose: The purpose of this trial is to investigate whether a microfluidics assay can detect trace amounts of residual leukemia and predict relapse in acute myeloid leukemia (AML) patients in remission who have undergone allogeneic stem cell transplantation (SCT) or Induction and Consolidation Chemotherapy (ICC) at the North Carolina Cancer Hospital (NCCH).

Procedures (methods): A total of 40 eligible subjects will be treated per standard of care with either SCT or induction and consolidation chemotherapy (ICC) based on the appropriate AML treatment paradigm for their disease. Peripheral blood (10 ml) for microfluidic chip analysis and possible Immune Monitoring Core Facility analysis will be collected along with routine lab draws prior to SCT. Patients in remission after SCT or those with confirmed remission by bone marrow biopsy after induction chemotherapy will be followed for 1 year; and peripheral blood (20 ml) will be collected to assess MRD by standard methods or by microfluidic chip analysis on a monthly basis. In addition, bone marrow biopsies will be performed at the end of consolidation (typically 5 months from remission), and at 1-year post remission in non-transplant patients. In transplanted patients, bone marrow biopsies will be collected at + 30 days, + 90 days, +180 days, and +360 days after SCT.

DETAILED DESCRIPTION:
An unmet need in the treatment of AML is earlier detection of potential relapse by monitoring MRD. The hope is that if clinicians can pinpoint when a patient's MRD starts towards a rapid expansion to relapse, preemptive therapies can be instituted earlier with the hope of eliciting improved outcomes. Current methods fall short of the ability to properly monitor MRD in individual patients. An ideal MRD assay would be easy to conduct, sensitive to low MRD levels and suitable for frequent analysis. A significant challenge for achieving this in AML is that unlike other leukemias, AML's interpatient heterogeneity is immense; and there is no characteristic genetic mutation or aberrant protein expression pattern for AML patients , thus hindering the broad applicability of polymerase chain reaction (PCR), fluorescence in-situ hypbridization (FISH) or multi-parameter flow cytometry (MFC) testing for MRD. Furthermore, AML relapse is rapid and it's been calculated that 42 day sampling intervals would be a minimum frequency needed to predict 75% of relapses during follow up after chemotherapy or SCT.

The microfluidics assay being evaluated in this study is relatively inexpensive, broadly applicable, as it identifies almost all (>90%) of AML cells, and easy to use. The microfluidic chip device is constructed with antibodies immobilized within the chip that can detect cell surface antigens commonly expressed on leukemic cells (ie, CD33, CD34, CD117, and CD123) directly in the peripheral blood without requiring preprocessing. The captured cells are then exposed to fluorescent antibodies targeting surface proteins that are aberrantly expressed on AML blasts (eg CD7, CD56 etc.), and fluorescence microscopy is used to identify captured cells that express an aberrant surface protein. The investigators have already completed a pilot study using this technology to monitor 5 AML patients after SCT. Because this assay required peripheral blood and not a bone marrow biopsy, 39 microfluidic tests could be carried out compared to only 8 PCR, MFC, FISH, and/or microscopy tests. Moreover, the frequent testing allowed us to observe signs of impending relapse earlier than the bone marrow biopsy-based test. The investigators plan to build on our findings in this trial and test the applicability of using the microfluidic assay for early signs of AML relapse. If successful, the microfluidic chip assay could be employed for serial MRD evaluations both in the post-SCT setting and in patients with AML undergoing conventional chemotherapy while providing a venue for the detailed management of a particular patient's AML including response to therapy and risk for disease recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥18 years of age) with newly diagnosed or suspected AML who are going to undergo stem cell transplant (SCT) or are being treated with induction and consolidation chemotherapy (ICC) at the NCCH are eligible. These subjects must provide written informed consent to participate.

   --For the purposes of this study, induction chemotherapy is any therapy intended to induce remission in AML patients that combines anthracycline/anthracenedione with cytarabine; or combinations of cytarabine at a dose of ≥1 g/m2/dose x ≥ 5 doses with a purine analogue. Liposomal combinations of anthracycline and cytarabine are also considered induction therapy. Subjects receiving investigational induction therapies will be eligible as long as the standard-of-care agents within the induction therapy fulfills criteria above.

   For the purposes of this study, specific choice of consolidation chemotherapy, or decision to pursue SCT in remission are not mandated prior to enrollment, as these decisions are not typically made until after induction chemotherapy has been given.
2. Subjects scheduled for SCT or ICC must have confirmed CD33-, CD34-, CD117- or CD123-positive disease to qualify for enrollment to undergo serial blood draws for assessment of MRD by microfluidic chip analysis.
3. Subjects may be enrolled after beginning induction chemotherapy, provided that sufficient AML blasts are available in the pre-treatment peripheral blood or bone marrow sample to confirm that the blasts express CD33, CD34, CD117 or CD123.

Exclusion Criteria:

1. Adult patients (≥18 years of age) with newly diagnosed or suspected AML who are scheduled to undergo SCT or ICC at the NCCH who do not provide written informed consent to participate are ineligible.
2. Patients who are receiving non-intense therapies for AML that do not contain anthracycline/anthracenedione or dual analog therapies. Such non-intense therapies include: DNA methyltransferase inhibitors (azacitidine/decitabine), combinations including DNA methyltransferase inhibitors, cytarabine monotherapy at doses below 1 g/m2 x 5, purine analog monotherapy or investigational therapies that are not combined with standard induction agents.
3. Subjects who test negative for the leukemic blasts surface antigens CD33, CD34, CD117, and CD123 are ineligible for inclusion to undergo serial blood draws for assessment of MRD by microfluidic chip analysis.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years of age) with newly diagnosed or suspected AML who are going to undergo stem cell transplant (SCT) or are being treated with induction and consolidation chemotherapy (ICC).
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2020-10-28 (Actual)

PRIMARY OUTCOMES:
Assessment of rising Minimal Residual Disease | The study will enroll 40 subjects with newly diagnosed or suspected AML or those who are transplant eligible. Subjects with confirmed remission after induction chemotherapy or after SCT will be followed for 1 year.
  The number of detected AML cells will be recorded for each obtained blood sample. An indicator of relapse is when the number of AML cells exceeds the threshold pre-specified before the study. The goal is to evaluate the sensitivity and specificity of the device against clinically confirmed relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Armistead, MD, Principal Investigator — UNC
Locations (1):
- UNC Lineberger, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No